CLINICAL TRIAL: NCT03992014
Title: A Two-period Study in Healthy Male Participants to Determine the Pharmacokinetics, Balance/Excretion, and Metabolism of [14C]-Linerixibat Following a Single Intravenous Radiolabeled Microtracer Dose (Concomitant With a Non-radiolabeled Oral Dose) and a Single Oral Radiolabeled Dose
Brief Title: Pharmacokinetics (PKs) and Metabolism of Radiolabelled Linerixibat
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205895
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Results first posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-05

CONDITIONS: Cholestasis
Keywords: [14C]-linerixibat; GSK2330672; Microtracer dose
MeSH Terms: conditions — Cholestasis

STUDY DESIGN:
Intervention Model Description: Subjects will receive linerixibat tablets concomitantly with [14C]-linerixibat IV infusion in treatment Period 1 and [14C]-linerixibat oral solution in treatment Period 2.
Masking Description: This will be an open-label study. Hence, there will be no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Linerixibat + [14C]-linerixibat (Experimental): Subjects will receive a single oral dose of linerixibat 90 milligram (mg) (2*45 mg) tablets concomitantly with [14C]-linerixibat 100 microgram (approximately 9.25 kilobecquerel; 250 nano curie) IV infusion for 3 hours, after an overnight fast that continues for 2 hours after the oral dose/start of IV infusion, small standard high-fat meal will be given on Day 1 in treatment Period 1; followed by a single oral dose of [14C]-linerixibat 90 mg (approximately 4.96 megabecquerel; 134.1 micro curie) solution on Day 1 in treatment Period 2. A wash out period of at least 13 days will be maintained between oral doses of treatment periods.
  Interventions: Drug: Linerixibat tablet; Drug: [14C]-linerixibat intravenous infusion; Drug: Linerixibat oral solution

INTERVENTIONS:
Drug: Linerixibat tablet — Linerixibat will be available as white to slightly colored film-coated round tablet to be administered as two tablets taken in the fasted state in the morning with 240 milliliter (mL) of room temperature water.
Drug: [14C]-linerixibat intravenous infusion — [14C]-linerixibat will be available as clear, colorless solution free from visible particulates to be administered 25 mL IV over 3 hours immediately after the oral dose.
Drug: Linerixibat oral solution — Linerixibat will be available as clear, colorless solution free from visible particulates to be administered 60 mL solution in the fasted state in the morning.

SUMMARY:
Absorption, metabolism and excretion of linerixibat have been studied in previous clinical trials. However, no dedicated clinical studies of drug absorption, metabolism, and excretion have been conducted for linerixibat. The purpose of this study is to determine the PK, balance/excretion, and metabolism of radiolabeled 14 Carbon [14C]-linerixibat following a single intravenous (IV) radiolabeled microtracer dose (concomitant with a non-radiolabeled oral dose) and a single oral radiolabeled dose. This is a single group, two period, single sequence, and mass balance study will enroll 6 healthy male subjects. Each subject will be involved in the study for up to 10 weeks which includes screening period, two treatment periods (treatment Periods 1 and 2), separated by about 7 days (at least 13 days between oral doses), and a follow-up visit 1-2 weeks after the last assessment in treatment Period 2.

ELIGIBILITY:
Inclusion Criteria

* Aged 30 to 55 years, inclusive, at the time of signing the informed consent.
* Healthy, as determined by the investigator or medically qualified designee, based on a medical evaluation including medical history, physical examination, vital signs, laboratory tests, and ECG. A subject with a clinical abnormality or laboratory parameter (i.e., outside the reference range for the population being studied), which is not specifically listed in the eligibility criteria, may be included only if the investigator agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* History of regular bowel movements (averaging one or more bowel movements per day).
* Non-smoker, or ex-smoker who hasn't regularly smoked for the 6 months before screening.
* Body weight of 50 kilogram and above, and body mass index (BMI) within the range 19.0 to 31.0 kilogram per square meter (kg/m^2) (inclusive).
* Male only. Subjects must agree to use contraception as follows: subjects with female partners of childbearing potential must agree to use a condom from the time of first dose of study intervention until 1 month after their last dose.
* Capable of giving signed informed consent.

Exclusion Criteria

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones). Subjects with a history of cholecystectomy must be excluded.
* Significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Any clinically relevant abnormality identified at the screening medical assessment (physical examination/medical history) clinical laboratory tests, or 12-lead ECG.
* Current episode, recent history, or chronic history of diarrhoea.
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Any current medical condition (example given [e.g.], psychiatric disorder, senility, dementia, or other condition), clinical or laboratory abnormality, or examination finding that the investigator considers would put the subjects at unacceptable risk, which may affect study compliance or prevent understanding of the aims or investigational procedures or possible consequences of the study.
* Regular use of known drugs of abuse or history of drug abuse or dependence within 6 months of the study.
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of >21 units. One unit is equivalent to 8 gram of alcohol: a glass (approximately 240 mL) of beer, 1 small glass (approximately 100 mL) of wine or 1 (approximately 25 mL) measure of spirits.
* History of or regular use of tobacco- or nicotine-containing products in the 6 months prior to screening.
* Past or intended use of over-the-counter or prescription medication, including analgesics (e.g., paracetamol), herbal medications, or grapefruit and Seville orange juices within 14 days prior to the first dose of study intervention until completion of the follow-up visit.
* Administration of any other Ileal bile acid transporter (IBAT) inhibitor in the 3 months prior to screening.
* Current enrolment in a clinical trial; recent participation in a clinical trial and has received an investigational product within 3 months before the first dose in the current study.
* Exposure to more than 4 new chemical entities within 12 months before the first dose in the current study.
* Participation in a clinical trial involving administration of 14C-labelled compound(s) within the last 12 months. A subjects previous effective dose will be reviewed by the medical investigator to ensure there is no risk of contamination/carryover into the current study.
* Received a total body radiation dose of greater than 10.0 millisievert (upper limit of International Commission on Radiological Protection [IRCP] category II) or exposure to significant radiation (e.g., serial x-ray or computed tomography [CT] scans, barium meal, etc.) in the 3 years before this study.
* Alanine transaminase (ALT) >1.5* upper limit of normal (ULN).
* Bilirubin >1.5*ULN (isolated bilirubin >1.5*ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* Presence of Hepatitis B surface antigen (HBsAg) at screening or positive Hepatitis C antibody test result at screening or within 3 months before the first dose of study intervention.
* Screening estimated glomerular filtration rate (eGFR) <45 milliliter per minute per 1.73 square meter (mL/min/1.73m^2) based on the Modification of Diet in Renal Disease (MDRD) Study equation.
* Positive pre-study drug/alcohol screen.
* Urinary cotinine levels indicative of smoking.
* Positive human immunodeficiency virus (HIV) antibody test.
* QT duration corrected for heart rate by Fridericia's formula >450 millisecond on ECG performed at Screening
* At screening or prior to the first dose, a supine blood pressure that is persistently higher than 140/90 millimeters of mercury (mmHg) taken in triplicate, unless deemed not clinically significant by the investigator.
* At screening or prior to the first dose, a supine mean heart rate outside the range of 40-100 beats per minute, unless deemed not clinically significant by the investigator.
* Has had an occupation which requires monitoring for radiation exposure, nuclear medicine procedures, or excessive x-rays within the past 12 months.
* Unable to refrain from consumption of prohibited food and drinks from 7 days before the first dose of study medication until the follow up visit.
* Loss of more than 400 mL blood during the 3 months before screening, e.g. as a blood donor, or plan to donate blood or blood products in the 3 months after the end of the trial.
* Unwillingness or inability to follow the procedures outlines in the protocol, including the use of the string bile collection device.
* History of sensitivity to linerixibat, or their components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline Medical Monitor, contraindicates their participation.

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only healthy male subjects will be enrolled in this study.
Enrollment: 6 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two-period, mass balance study in healthy male participants to assess the pharmacokinetics (PK), excretion and metabolism of Linerixibat. The study was conducted at a single center in the United Kingdom.
Pre-assignment Details: A total of 10 participants were screened of which 4 failed screening and 6 participants were enrolled in the study. The study had 2 treatment periods (each of 8 days) with a washout of 7 days. All participants were followed-up at Day 34.
Groups:
- Linerixibat Tab+[14C]Linerixibat IV/[14C] Linerixibat Oral Sol: Participants were administered a single oral dose of 90 milligram (mg) linerixibat (two tablets [tab] of 45 mg each) in fasted state followed by an intravenous (IV) infusion of 100 micrograms (μg) radiolabeled [14C]-linerixibat infused over 3 hours on Day 1 of treatment period 1. Participants received 60 milliliter (mL) of 90 mg [14C]-linerixibat oral solution (sol) in the fasted state on Day 1 of treatment period 2. The treatment periods were separated by a washout period of about 7 days (at least 13 days between oral doses). All participants were followed-up at Day 34.
Period: Treatment Period 1 (8 Days)
Arm/Group | Linerixibat Tab+[14C]Linerixibat IV/[14C] Linerixibat Oral Sol
Started | 6
Completed | 6
Not Completed | 0
Period: Washout Period (7 Days)
Arm/Group | Linerixibat Tab+[14C]Linerixibat IV/[14C] Linerixibat Oral Sol
Started | 6
Completed | 6
Not Completed | 0
Period: Treatment Period 2 (8 Days)
Arm/Group | Linerixibat Tab+[14C]Linerixibat IV/[14C] Linerixibat Oral Sol
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Linerixibat Tab+[14C]Linerixibat IV/[14C] Linerixibat Oral Sol
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 2
  White - White/Caucasian/European Heritage | 4

OUTCOME MEASURES:

1. Primary Outcome: Period 1: Area Under the Concentration-time Curve (AUC) From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC[0-inf]) of Linerixibat and [14C]-Linerixibat Following Oral Dose of Linerixibat and IV Dose of [14C]-Linerixibat
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population comprised of all participants in the Safety Population (all participants who took atleast one dose of study treatment) who had at least 1 non-missing PK assessment. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram per milliliter
Groups:
- Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV: Eligible participants received 25 mL of intravenous (IV) radiolabelled [14C]-Linerixibat 100 microgram (μg) infused over 3 hours immediately after the Linerixibat 90 mg (two 45 mg) tablets orally in fasted state on Day 1 of treatment period 1.
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV
Number analyzed (Participants) | 6
Hours*picogram per milliliter
  Linerixibat 90 mg oral tablets | 1554 (25.8)
  [14C] Linerixibat 100 μg IV | 1570 (26.7)

2. Primary Outcome: Period 2: AUC(0-inf) of [14C]-Linerixibat Following Administration of Oral Dose of [14C]-Linerixibat Solution
Description: as for outcome 1
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram per milliliter
Groups:
- [14C]-Linerixibat 90 Milligram Oral Solution: Participants received single 60 mL oral solution of 90 mg [14C]-Linerixibat on Day 1 of treatment period 2 in fasted state
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 3
Hours*picogram per milliliter | 1634 (95.3)

3. Primary Outcome: Period 1: AUC From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC[0-t]) of Linerixibat and [14C]-Linerixibat Following Oral Dose of Linerixibat and IV Dose of [14C]-Linerixibat
Description: as for outcome 1
Time Frame: as for outcome 1
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram per milliliter
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV
Number analyzed (Participants) | 6
Hours*picogram per milliliter
  Linerixibat 90 mg oral tablets | 749 (125)
  [14C] Linerixibat 100 μg IV | 1560 (26.8)

4. Primary Outcome: Period 2: AUC(0-t) of [14C]-Linerixibat Following Administration of Oral Dose of [14C] Linerixibat Solution
Description: Blood samples were collected at indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram per milliliter
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Hours*picogram per milliliter | 1044 (79.4)

5. Primary Outcome: Period 1: Maximum Observed Concentration (Cmax) of Linerixibat and [14C]-Linerixibat Following Oral Dose of Linerixibat and IV Dose of [14C]-Linerixibat
Description: as for outcome 4
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV
Number analyzed (Participants) | 6
Picogram per milliliter
  Linerixibat 90 mg oral tablets | 120 (108)
  [14C] Linerixibat 100 μg IV | 638 (27.3)

6. Primary Outcome: Period 2: Cmax of [14C]-Linerixibat Following Administration of Oral Dose of [14C] Linerixibat Solution
Description: as for outcome 4
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Picogram per milliliter | 158 (270)

7. Primary Outcome: Period 1: Time of Occurrence of Cmax (Tmax) of Linerixibat and [14C]-Linerixibat Following Oral Dose of Linerixibat and IV Dose of [14C]-Linerixibat
Description: as for outcome 4
Time Frame: as for outcome 1
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV
Number analyzed (Participants) | 6
Hours
  Linerixibat 90 mg oral tablets | 2.25 [0.500 to 5.50]
  [14C] Linerixibat 100 μg IV | 1.49 [0.983 to 2.50]

8. Primary Outcome: Period 2: Tmax of [14C]-Linerixibat Following Administration of Oral Dose of [14C] Linerixibat Solution
Description: as for outcome 4
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Hours | 7.50 [2.00 to 48.1]

9. Primary Outcome: Period 1: Terminal Phase Half-Life (t1/2) of Linerixibat and [14C]-Linerixibat Following Oral Dose of Linerixibat and IV Dose of [14C]-Linerixibat
Description: as for outcome 1
Time Frame: as for outcome 1
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV
Number analyzed (Participants) | 6
Hours
  Linerixibat 90 mg oral tablets | 6.76 (124)
  [14C] Linerixibat 100 μg IV | 0.828 (18.3)

10. Primary Outcome: Period 2: t1/2 of [14C]-Linerixibat Following Administration of Oral Dose of [14C] Linerixibat Solution
Description: as for outcome 4
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 3
Hours | 6.25 (64.3)

11. Primary Outcome: Period 1: AUC(0-inf) of Total Radioactivity Following IV Dose of [14C]-Linerixibat
Description: Blood samples were collected at the indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. Not applicable (NA) indicates geometric coefficient of variation could not be calculated as a single participant was analyzed.
Time Frame: as for outcome 1
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram equivalent per milliliter
Groups:
- [14C]-Linerixibat 100 Microgram Intravenous Infusion: Participants received single 25 mL IV dose of radiolabelled [14C]-Linerixibat 100 μg infused over 3 hours on Day 1 of treatment period 1.
Arm/Group | [14C]-Linerixibat 100 Microgram Intravenous Infusion
Number analyzed (Participants) | 1
Hours*picogram equivalent per milliliter | 2300 (NA) — Not applicable (NA) indicates geometric coefficient of variation could not be calculated as a single participant was analyzed.

12. Primary Outcome: Period 2: AUC(0-inf) of Total Radioactivity Following Administration of Oral Dose of [14C]-Linerixibat Solution
Description: as for outcome 1
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram equivalent per milliliter
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Hours*picogram equivalent per milliliter | 94740 (8.17)

13. Primary Outcome: Period 1: AUC(0-t) of Total Radioactivity Following IV Dose of [14C]-Linerixibat
Description: as for outcome 1
Time Frame: as for outcome 1
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram equivalent per milliliter
Arm/Group | [14C]-Linerixibat 100 Microgram Intravenous Infusion
Number analyzed (Participants) | 6
Hours*picogram equivalent per milliliter | 1903 (22.3)

14. Primary Outcome: Period 2: AUC(0-t) of Total Radioactivity Following Administration of Oral Dose of [14C] Linerixibat Solution
Description: as for outcome 4
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram equivalent per milliliter
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Hours*picogram equivalent per milliliter | 67533 (11.3)

15. Primary Outcome: Period 1: Cmax of Total Radioactivity Following IV Dose of [14C]-Linerixibat
Description: as for outcome 4
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram equivalent per milliliter
Arm/Group | [14C]-Linerixibat 100 Microgram Intravenous Infusion
Number analyzed (Participants) | 6
Picogram equivalent per milliliter | 738 (23.6)

16. Primary Outcome: Period 2: Cmax of Total Radioactivity Following Administration of Oral Dose of [14C] Linerixibat Solution
Description: as for outcome 4
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram equivalent per milliliter
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Picogram equivalent per milliliter | 2784 (14.3)

17. Primary Outcome: Period 1: Tmax of Total Radioactivity Following IV Dose of [14C]-Linerixibat
Description: as for outcome 4
Time Frame: as for outcome 1
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | [14C]-Linerixibat 100 Microgram Intravenous Infusion
Number analyzed (Participants) | 6
Hours | 1.49 [0.983 to 2.00]

18. Primary Outcome: Period 2: Tmax of Total Radioactivity Following Administration of Oral Dose of [14C] Linerixibat Solution
Description: as for outcome 4
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Hours | 0.50 [0.500 to 1.00]

19. Primary Outcome: Period 1: t1/2 of [14C]-Linerixibat for Total Radioactivity Following IV Dose of [14C]-Linerixibat
Description: as for outcome 1
Time Frame: as for outcome 1
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | [14C]-Linerixibat 100 Microgram Intravenous Infusion
Number analyzed (Participants) | 1
Hours | 0.733 (NA) — NA indicates geometric coefficient of variation could not be calculated as a single participant was analyzed.

20. Primary Outcome: Period 2: t1/2 of [14C]-Linerixibat for Total Radioactivity Following Administration of Oral Dose of [14C] Linerixibat Solution
Description: as for outcome 4
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144 and 168 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Hours | 98.3 (13.7)

21. Primary Outcome: Period 1: Volume of Distribution at Steady State (Vss) of [14C]-Linerixibat Following Administration of IV Dose of [14C]-Linerixibat
Description: as for outcome 4
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter
Arm/Group | [14C]-Linerixibat 100 Microgram Intravenous Infusion
Number analyzed (Participants) | 6
Milliliter | 16340 (35.7)

22. Primary Outcome: Period 1: Total Plasma Clearance (CL) of [14C]-Linerixibat Following Administration of IV Dose of [14C]-Linerixibat
Description: as for outcome 1
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters per minute
Arm/Group | [14C]-Linerixibat 100 Microgram Intravenous Infusion
Number analyzed (Participants) | 6
Milliliters per minute | 1032 (27.3)

23. Primary Outcome: Period 1: Hepatic Clearance (CLh) of [14C]-Linerixibat Following Administration of IV Dose of [14C]-Linerixibat
Description: Blood samples were collected at indicated time points for PK analysis. PK parameters were calculated by standard non-compartmental analysis. Hepatic clearance was calculated as total plasma IV clearance minus renal clearance.
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters per minute
Arm/Group | [14C]-Linerixibat 100 Microgram Intravenous Infusion
Number analyzed (Participants) | 6
Milliliters per minute | 867 (26.4)

24. Primary Outcome: Period 1: Absolute Oral Bioavailability (F) of Linerixibat Following Administration of Oral Dose of Linerixibat and IV Dose of [14C]-Linerixibat
Description: Blood samples were collected at indicated time points for PK analysis. Absolute bioavailability is the amount of drug from a formulation that reaches the systemic circulation relative to an IV dose. It is expressed as percentage bioavailability, which is calculated by ratio of AUC(oral)/Dose(oral) with AUC(IV)/Dose(IV) multiplied by 100.
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage bioavailability
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV
Number analyzed (Participants) | 6
Percentage bioavailability | 0.0517 (120)

25. Primary Outcome: Period 1: Percentage of Drug Escaping First-pass Hepatic Clearance (Fh) of Linerixibat Following Administration of Oral Dose of Linerixibat and IV Dose of [14C]-Linerixibat
Description: Blood samples were collected from participants at indicated time points. Fh was expressed as percentage and was calculated as: 1 minus hepatic extraction ratio multiplied by 100. Hepatic extraction ratio=hepatic blood clearance (milliliters per minute)/hepatic blood flow (milliliters per minute).
Time Frame: as for outcome 1
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of drug escaped
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV
Number analyzed (Participants) | 5
Percentage of drug escaped | 24.4 (68.4)

26. Primary Outcome: Period 1: Percentage of Drug Absorbed (Fa) for Linerixibat Following Administration of Oral Dose of Linerixibat and IV Dose of [14C]-Linerixibat
Description: Blood samples were collected from participants at indicated time points. Fa was expressed as percentage which was calculated as ratio of oral bioavailability and Fh multiplied by 100.
Time Frame: as for outcome 1
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of drug absorbed
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV
Number analyzed (Participants) | 5
Percentage of drug absorbed | 0.167 (73.7)

27. Primary Outcome: Period 1: Summary of Mean Cumulative Total Recovery (Percentage Excreted) in Urine Following Administration of IV Dose of [14C]-Linerixibat.
Description: Urine samples were collected at indicated time points and total radioactivity measurement was done using Liquid Scintillation counting (LSC). Percentage of radioactive dose excreted in urine was calculated as (amount excreted in urine divided by administered radioactivity dose) multiplied by 100.
Time Frame: 0-24, 0-48, 0-72, 0-96, 0-120, 0-144 and 0-168 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Percentage dose
Arm/Group | [14C]-Linerixibat 100 Microgram Intravenous Infusion
Number analyzed (Participants) | 6
Percentage dose
  0-24 Hours | 16.4 (2.8)
  0-48 Hours | 16.4 (2.8)
  0-72 Hours | 16.5 (2.8)
  0-96 Hours | 16.5 (2.8)
  0-120 Hours | 16.5 (2.8)
  0-144 Hours | 16.5 (2.8)
  0-168 Hours | 16.5 (2.8)

28. Primary Outcome: Period 2: Summary of Mean Cumulative Total Recovery (Percentage Excreted) in Urine Following Administration of Oral Dose of [14C]-Linerixibat
Description: Urine samples were collected at indicated time points and total radioactivity measurement was done using LSC. Percentage of radioactive dose excreted in urine was calculated as (amount excreted in urine divided by administered radioactivity dose) multiplied by 100.
Time Frame: 0-24, 0-48, 0-72, 0-96, 0-120, 0-144 and 0-168 hours post-dose
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Percentage dose
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Percentage dose
  0-24 Hours | 0.04 (0.03)
  0-48 Hours | 0.04 (0.03)
  0-72 Hours | 0.04 (0.03)
  0-96 Hours | 0.04 (0.03)
  0-120 Hours | 0.04 (0.03)
  0-144 Hours | 0.04 (0.03)
  0-168 Hours | 0.04 (0.03)

29. Primary Outcome: Period 1: Summary of Mean Cumulative Total Recovery (Percentage Excreted) in Feces Following Administration of IV Dose of [14C]-Linerixibat
Description: Feces samples were collected at indicated time points and total radioactivity measurement was done using LSC. Percentage of radioactive dose excreted was calculated as (amount excreted in feces homogenate divided by administered radioactivity dose) multiplied by 100.
Time Frame: 0-24, 0-48, 0-72, 0-96, 0-120, 0-144 and 0-168 hours post-dose
Population: PK Population
Measure: Mean (Standard Deviation); unit: Percentage dose
Arm/Group | [14C]-Linerixibat 100 Microgram Intravenous Infusion
Number analyzed (Participants) | 6
Percentage dose
  0-24 Hours | 33.4 (19.4)
  0-48 Hours | 43.6 (18.8)
  0-72 Hours | 61.3 (7.5)
  0-96 Hours | 67.8 (6.3)
  0-120 Hours | 68.8 (6.3)
  0-144 Hours | 69.1 (6.3)
  0-168 Hours | 69.2 (6.3)

30. Primary Outcome: Period 2: Summary of Mean Cumulative Total Recovery (Percentage Excreted) in Feces Following Administration of Oral Dose of [14C]-Linerixibat
Description: as for outcome 29
Time Frame: 0-24, 0-48, 0-72, 0-96, 0-120, 0-144 and 0-168 hours post-dose
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage dose
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 5
Percentage dose
  0-24 Hours | 41.2 (46.5)
  0-48 Hours | 64.4 (40.6)
  0-72 Hours | 84.4 (15.7)
  0-96 Hours | 93.2 (7.8)
  0-120 Hours | 96.3 (2.9)
  0-144 Hours | 97.0 (2.7)
  0-168 Hours | 97.1 (2.7)

31. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study treatment. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgement.
Time Frame: Up to 34 days
Population: Safety Population comprised of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6 | 6
Participants
  Any AEs | 3 | 3
  Any SAEs | 0 | 0

32. Secondary Outcome: Number of Participants With Worst Case Hematology Results Relative to Normal Range
Description: Blood samples were collected to analyze the following hematology parameters; Basophils, Eosinophils, Erythrocytes mean corpuscular volume (MCV), Erythrocytes mean corpuscular hemoglobin (MCH), Erythrocytes, Hematocrit (HCT), Hemoglobin (Hb), Leukocytes, Lymphocytes, Monocytes, Neutrophils, Platelets, Reticulocytes and Reticulocytes/Erythrocytes. Participants were counted in the worst case category if their value changes to (low, normal or high), unless there was no change in their category. Participants whose laboratory value category was unchanged (e.g. High to High), or whose value became normal, were recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Up to 34 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6 | 6
Participants
  Basophils, To low | 0 | 0
  Basophils, To normal or no change | 6 | 6
  Basophils, To high | 0 | 0
  Eosinophils, To low | 0 | 0
  Eosinophils, To normal or no change | 6 | 6
  Eosinophils, To high | 0 | 0
  MCV, To low | 0 | 0
  MCV, To normal or no change | 6 | 6
  MCV, To high | 0 | 0
  MCH, To low | 0 | 1
  MCH, To normal or no change | 6 | 5
  MCH, To high | 0 | 0
  Erythrocytes, To low | 0 | 0
  Erythrocytes, To normal or no change | 6 | 6
  Erythrocytes, To high | 0 | 0
  HCT, To low | 0 | 0
  HCT, To normal or no change | 6 | 6
  HCT, To high | 0 | 0
  Hb, To low | 0 | 0
  Hb, To normal or no change | 6 | 6
  Hb, To high | 0 | 0
  Leukocytes, To low | 0 | 1
  Leukocytes, To normal or no change | 6 | 5
  Leukocytes, To high | 0 | 0
  Lymphocytes, To low | 0 | 1
  Lymphocytes, To normal or no change | 6 | 5
  Lymphocytes, To high | 0 | 0
  Monocytes, To low | 0 | 0
  Monocytes, To normal or no change | 6 | 6
  Monocytes, To high | 0 | 0
  Neutrophils, To low | 0 | 0
  Neutrophils, To normal or no change | 6 | 6
  Neutrophils, To high | 0 | 0
  Platelets, To low | 0 | 0
  Platelets, To normal or no change | 6 | 6
  Platelets, To high | 0 | 0
  Reticulocytes, To low | 0 | 0
  Reticulocytes, To normal or no change | 6 | 6
  Reticulocytes, To high | 0 | 0
  Reticulocytes/Erythrocytes, To low | 0 | 0
  Reticulocytes/Erythrocyte, To normal or no change | 6 | 6
  Reticulocytes/Erythrocytes, To high | 0 | 0

33. Secondary Outcome: Number of Participants With Worst Case Chemistry Results Relative to Normal Range
Description: Blood samples were collected to analyze the following clinical chemistry parameters; alanine aminotransferase (ALT), albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), bilirubin, calcium, chloride, cholesterol, creatinine, direct bilirubin, globulin, glucose, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, phosphate, potassium, protein, sodium, triglycerides, urate and urea. Participants were counted in the worst case category if their value changes to (low, normal or high), unless there was no change in their category. Participants whose laboratory value category was unchanged (e.g. High to High), or whose value became normal, were recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100%.
Time Frame: Up to 34 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6 | 6
Participants
  ALT, To low | 0 | 0
  ALT, To normal or no change | 6 | 6
  ALT, To high | 0 | 0
  Albumin, To low | 0 | 0
  Albumin, To normal or no change | 6 | 6
  Albumin, To high | 0 | 0
  ALP, To low | 0 | 0
  ALP, To normal or no change | 6 | 6
  ALP, To high | 0 | 0
  AST, To low | 0 | 0
  AST, To normal or no change | 6 | 6
  AST, To high | 0 | 0
  Bilirubin, To low | 0 | 0
  Bilirubin, To normal or no change | 6 | 6
  Bilirubin, To high | 0 | 0
  Calcium, To low | 0 | 0
  Calcium, To normal or no change | 6 | 6
  Calcium, To high | 0 | 0
  Chloride, To low | 0 | 0
  Chloride, To normal or no change | 6 | 6
  Chloride, To high | 0 | 0
  Cholesterol, To low | 0 | 0
  Cholesterol, To normal or no change | 6 | 6
  Cholesterol, To high | 0 | 0
  Creatinine, To low | 0 | 0
  Creatinine, To normal or no change | 6 | 6
  Creatinine, To high | 0 | 0
  Direct Bilirubin, To low | 0 | 0
  Direct Bilirubin, To normal or no change | 6 | 6
  Direct Bilirubin, To high | 0 | 0
  Globulin, To low | 0 | 0
  Globulin, To normal or no change | 6 | 6
  Globulin, To high | 0 | 0
  Glucose, To low | 0 | 0
  Glucose, To normal or no change | 6 | 6
  Glucose, To high | 0 | 0
  HDL Cholesterol, To low | 0 | 0
  HDL Cholesterol, To normal or no change | 6 | 5
  HDL Cholesterol, To high | 0 | 1
  LDL Cholesterol, To low | 0 | 0
  LDL Cholesterol, To normal or no change | 3 | 5
  LDL Cholesterol, To high | 3 | 1
  Phosphate, To low | 0 | 0
  Phosphate, To normal or no change | 6 | 6
  Phosphate, To high | 0 | 0
  Potassium, To low | 0 | 0
  Potassium, To normal or no change | 6 | 6
  Potassium, To high | 0 | 0
  Protein, To low | 0 | 0
  Protein, To normal or no change | 6 | 6
  Protein, To high | 0 | 0
  Sodium, To low | 0 | 0
  Sodium, To normal or no change | 6 | 6
  Sodium, To high | 0 | 0
  Triglycerides, To low | 0 | 0
  Triglycerides, To normal or no change | 6 | 6
  Triglycerides, To high | 0 | 0
  Urate, To low | 0 | 0
  Urate, To normal or no change | 6 | 6
  Urate, To high | 0 | 0
  Urea, To low | 0 | 0
  Urea, To normal or no change | 6 | 6
  Urea, To high | 0 | 0

34. Secondary Outcome: Number of Participants With Abnormal Urinalysis Results by Dipstick Method
Description: Urine samples were collected to assess urine glucose, urine protein, urine blood, urine ketones, urine bilirubin, urine urobilinogen, urine nitrite and urine leukocyte esterase by dipstick test. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameter can be read as negative (-) and positive (+) indicating proportional concentrations in the urine sample. Number of participants who had abnormal findings in any of these urinalysis parameters are presented.
Time Frame: Up to 34 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

35. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Findings for Electrocardiogram (ECG) Parameters
Description: Full 12-lead ECGs were recorded with the participants in a supine position. 12-lead ECGs were obtained using an automated ECG machine that measured PR, QRS, QT and QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals and calculated heart rate. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. The number of participants with clinically significant abnormal findings for ECG parameters at worst-case post Baseline are presented.
Time Frame: Up to 34 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

36. Secondary Outcome: Period 1: Change From Baseline in Diastolic Blood Pressure (DBP) at Indicated Time-points
Description: DBP was measured in a semi-recumbent position after 5 minutes of rest for the participant. Mean of the triplicate pre-dose assessments on Day 1 of treatment period 1 was considered as Baseline value. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline, Day 1 (4 Hours) and Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV
Number analyzed (Participants) | 6
Millimeters of mercury
  Day 1 (4 Hours) | -1.2 (4.11)
  Day 8 | 2.0 (8.81)

37. Secondary Outcome: Period 2: Change From Baseline in DBP at Indicated Time-points
Description: as for outcome 36
Time Frame: Baseline, Day 1 (4 Hours) and Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Millimeters of mercury
  Day 1 (4 Hours) | -2.4 (7.27)
  Day 8 | 2.1 (6.56)

38. Secondary Outcome: Change From Baseline in DBP at Follow-up Visit (Day 34)
Description: as for outcome 36
Time Frame: Baseline and Day 34 (post Day 1 of Period 1 dosing)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Millimeters of mercury | 1.2 (6.66)

39. Secondary Outcome: Period 1: Change From Baseline in Pulse Rate at Indicated Time-points
Description: Pulse rate was measured in a semi-recumbent position after 5 minutes of rest for the participant. Mean of the triplicate pre-dose assessments on Day 1 of treatment period 1 was considered as Baseline value. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value
Time Frame: Baseline, Day 1 (4 Hours) and Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV
Number analyzed (Participants) | 6
Beats per minute
  Day 1 (4 Hours) | 1.3 (4.20)
  Day 8 | 1.9 (4.02)

40. Secondary Outcome: Period 2: Change From Baseline in Pulse Rate at Indicated Time-points
Description: as for outcome 39
Time Frame: Baseline, Day 1 (4 Hours) and Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Beats per minute
  Day 1 (4 Hours) | -0.6 (4.20)
  Day 8 | 1.3 (2.60)

41. Secondary Outcome: Change From Baseline in Pulse Rate at Follow-up Visit (Day 34)
Description: as for outcome 39
Time Frame: Baseline and Day 34 (post Day 1 of Period 1 dosing)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Beats per minute | 2.8 (7.79)

42. Secondary Outcome: Period 1: Change From Baseline in Systolic Blood Pressure (SBP) at Indicated Time-points
Description: SBP was measured in a semi-recumbent position after 5 minutes of rest for the participant. Mean of the triplicate pre-dose assessments on Day 1 of treatment period 1 was considered as Baseline value. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value
Time Frame: Baseline, Day 1 (4 Hours) and Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV
Number analyzed (Participants) | 6
Millimeters of mercury
  Day 1 (4 Hours) | 5.2 (11.16)
  Day 8 | 6.6 (7.68)

43. Secondary Outcome: Period 2: Change From Baseline in SBP at Indicated Time-points
Description: as for outcome 42
Time Frame: Baseline, Day 1 (4 Hours) and Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Millimeters of mercury
  Day 1 (4 Hours) | -1.1 (8.73)
  Day 8 | 6.5 (6.39)

44. Secondary Outcome: Change From Baseline in SBP at Follow-up Visit (Day 34)
Description: as for outcome 42
Time Frame: Baseline and Day 34 (post Day 1 of Period 1 dosing)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Millimeters of mercury | 2.4 (8.96)

45. Secondary Outcome: Period 1: Change From Baseline in Respiratory Rate at Indicated Time-points
Description: Respiratory rate was measured in a semi-recumbent position after 5 minutes of rest for the participant. Mean of the triplicate pre-dose assessments on Day 1 of treatment period 1 was considered as Baseline value. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value
Time Frame: Baseline, Day 1 (4 Hours) and Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV
Number analyzed (Participants) | 6
Breaths per minute
  Day 1 (4 Hours) | 0.0 (2.19)
  Day 8 | 1.0 (4.15)

46. Secondary Outcome: Period 2: Change From Baseline in Respiratory Rate at Indicated Time-points
Description: as for outcome 45
Time Frame: Baseline, Day 1 (4 Hours) and Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Breaths per minute
  Day 1 (4 Hours) | -0.7 (1.63)
  Day 8 | -0.7 (2.73)

47. Secondary Outcome: Change From Baseline in Respiratory Rate at Follow-up Visit (Day 34)
Description: as for outcome 45
Time Frame: Baseline and Day 34 (post Day 1 of Period 1 dosing)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Breaths per minute | -1.7 (3.67)

48. Secondary Outcome: Period 1: Change From Baseline in Tympanic Membrane Temperature at Indicated Time-points
Description: Tympanic membrane temperature was measured in a semi-recumbent position after 5 minutes of rest for the participant. Mean of the triplicate pre-dose assessments on Day 1 of treatment period 1 was considered as Baseline value. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline, Day 1 (4 Hours) and Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV
Number analyzed (Participants) | 6
Degree Celsius
  Day 1 (4 Hours) | 0.4 (0.37)
  Day 8 | -0.4 (0.63)

49. Secondary Outcome: Period 2: Change From Baseline in Tympanic Membrane Temperature at Indicated Time-points
Description: as for outcome 48
Time Frame: Baseline, Day 1 (4 Hours) and Day 8
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Degree Celsius
  Day 1 (4 Hours) | 0.2 (0.58)
  Day 8 | -0.4 (0.56)

50. Secondary Outcome: Change From Baseline in Tympanic Membrane Temperature at Follow-up Visit (Day 34)
Description: as for outcome 48
Time Frame: Baseline and Day 34 (post Day 1 of Period 1 dosing)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | [14C]-Linerixibat 90 Milligram Oral Solution
Number analyzed (Participants) | 6
Degree Celsius | 0.3 (0.37)

ADVERSE EVENTS:
Time Frame: SAEs and non-serious AEs were collected from the start of study treatment up to Day 34.
Description: SAEs and Non-SAEs were reported for the Safety Population which comprised of all participants who received at least one dose of study treatment
Arm/Group | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV | [14C]-Linerixibat 90 Milligram Oral Solution
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linerixibat 90 mg Oral Tablets + [14C] Linerixibat 100 μg IV (N=6) | [14C]-Linerixibat 90 Milligram Oral Solution (N=6)
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT03992014/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT03992014/SAP_001.pdf